CLINICAL TRIAL: NCT03644251
Title: FLO Injection for Discogenic Pain
Brief Title: FLO for Discogenic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Site Ceased all Business Operations
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLARIX-CS003
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Discogenic Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AMUC Dosage 1 (Experimental): 25mg amniotic and umbilical cord matrix
  Interventions: Other: amniotic and umbilical cord matrix
- AMUC Dosage 2 (Experimental): 50mg amniotic and umbilical cord matrix
  Interventions: Other: amniotic and umbilical cord matrix
- AMUC Dosage 3 (Experimental): 100mg amniotic and umbilical cord matrix
  Interventions: Other: amniotic and umbilical cord matrix

INTERVENTIONS:
Other: amniotic and umbilical cord matrix — Cryopreserved human amniotic and umbilical cord product derived from donated human placental tissue following healthy, live, caesarian section, full-term births after determination of donor eligibility and placenta suitability.

SUMMARY:
Discogenic pain is pain originating from a damaged vertebral disc and be caused by inflammation, dehydration of the nucleus pulposus, decreased disc height, annular tears and impaired mechanical function of the disc.Non-operative treatment may include traction, steroid therapy, methylene blue injection and ablative therapy. However, there are few high quality studies evaluating these treatments for reducing discogenic low back pain and most clinical trials failed to detect significant differences between treatments and placebo therapies. Hence, there remains an unmet clinical need.

ELIGIBILITY:
Inclusion Criteria:

* subject (male or female) is at least 18 to 70 years of age
* diagnosed with single level discogenic back pain confirmed by MRI and positive discography per Spine Interventional Society Guidelines
* Diagnosis of disc degeneration with Pfirrmann score of 1-3
* Subject has failed at least six months of conservative care
* Subject is symptomatic with axial lower back pain greater than lower limb pain at the intensity of >6/10 concordant or partially concordant
* The subject is able to comply with all post-operative standard of care and follow instructions.

Exclusion Criteria:

* Subjects has significant disc protrusion, severe lumbar spinal stenosis, spine tumor, severe disc degeneration, or Sacroiliac (SI) joint syndrome
* Subject had previous surgery at the disc level
* Patient has previously received injection of FLO within 3 months of screening
* The subject is unable to comply with follow-up or not appropriate for inclusion based on investigator decision

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Change in patient back pain determined by visual analog scale | 3 months
  0 to 100mm, 100mm worst pain

SECONDARY OUTCOMES:
Change in quality of life determined by SF-36 | 3 and 6 months
  Short FormHealth Survey to evaluate quality of life across eight scales
Change in patient back pain determined by visual analog scale | 6 months
  0 to 100mm, 100mm worst pain
Change in Oswestry Disability Index | 3 and 6 months
  0 to 50, higher the percentile, the worse the perceived lower back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Laser Spine Institute, Tampa, Florida, United States